CLINICAL TRIAL: NCT00004342
Title: International Registry for Severe Chronic Neutropenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, David Chandler Dale, Professor of Medicine, University of Washington
Other Study IDs: 199/11901; UW-730
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Neutropenia
Keywords: chronic neutropenia; disease-related problem/condition; hematologic disorders; neutropenia; rare disease; severe chronic neutropenia
MeSH Terms: conditions — Neutropenia; Hematologic Diseases; Rare Diseases; Neutropenia, severe chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, Bone marrow, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adult Neutropenic Subject: Adult subjects with diagnosis of severe chronic neutropenia
- Minor Neutropenic Subject: Children under 18 years of age who are diagnosed with severe chronic neutropenia
- Parent of Minor Neutropenic Subjects: Parent of minor subjects (i.e., children under 18 years of age) who are diagnosed with severe chronic neutropenia

SUMMARY:
OBJECTIVES: I. Document the clinical course of severe chronic neutropenia (SCN).

II. Monitor and assess long term safety of primary treatment in SCN patients in the United States, Canada, Europe, and Australia.

III. Study the incidence and outcome of adverse events such as osteoporosis, splenomegaly, cytogenetic abnormalities, myelodysplastic syndrome, and leukemia.

IV. Evaluate growth and development and hematologic parameters. V. Monitor for clinically significant changes in primary treatment response over time.

VI. Establish a physician network to increase the understanding of SCN. VII. Establish a demographic database to allow for future research.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients are treated by the referring physician as medically indicated. Clinical data are collected at baseline and then every 6 months.

ELIGIBILITY:
Inclusion Criteria - Subjects are eligible for enrollment if they meet the following criteria:

1. A confirmed diagnosis of severe chronic neutropenia based on documented absolute neutrophil counts of less than 0.5x109/L on at least three occasions in the three months prior to enrollment.
2. For subjects with presumed cyclic neutropenia, documentation of at least two neutrophil cycles is preferred. Documentation should include the nadirs with neutrophil counts of less than 200 followed by a clear increase in the counts generally to at least 500 to 1000 followed by a second nadir, usually expected to occur at about three weeks after the first nadir, i.e., cycling with a three week periodicity. Documentation with at least six weeks of counts and two expected nadirs is preferred.

   Cases not showing clear oscillations will be categorized as congenital (if neutropenia or neutropenic complications appear to have occurred from birth) or idiopathic (if all symptoms in evidence point to an acquired disorder occurring after the first year of life).
3. Bone marrow aspiration consistent with the diagnosis of congenital, cyclic or idiopathic neutropenia. In all of these conditions, it is expected that the marrow aspirate evaluation at the time of neutropenia will show a deficiency of mature neutrophils. An exception is myelokathexis, a condition with large accumulations of neutrophils with pycnotic nuclei in the marrow. Bone marrow aspirates may show some dyspoiesis of the neutrophil lineage, but abnormalities of erythropoiesis or platelet formation are, in general, inconsistent with the diagnosis of SCN.
4. Normal cytogenetic evaluation. The only exception being cases of well documented severe congenital neutropenia with preferably previously documented normal cytogenetic evaluation will now be enrolled in the Registry at the time of evolution to leukemia.
5. History of recurrent infections (i.e., severe mouth ulcers, gingivitis and sinusitis).
6. Age greater than three months.
7. Independent of hematological parameters, subjects with the following diagnoses may be included: Shwachman-Diamond syndrome (SDS), glycogen storage disease type 1b (GSD1b), Barth syndrome, and Cohen's syndrome.
8. Subjects with moderately severe chronic neutropenia (i.e., ANC less than 1.0x109/L) and recurrent severe infections (i.e., deep tissue infections of subcutaneous areas, lungs, liver, etc.).
9. Immune neutropenia with positive anti-neutrophil antibodies meeting criteria in 1, 3, 5 and 6.
10. All SCN subjects originally enrolled in Amgen-sponsored SCN studies.

Exclusion Criteria

1. Neutropenia known to be drug induced
2. Primary myelodysplasia
3. Primary leukemia
4. Aplastic anemia
5. Known HIV disease
6. Systemic autoimmune diseases such as rheumatoid arthritis or systemic lupus erythematosus
7. Chemotherapy-induced neutropenia (within the last 5 years)

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with severe chronic neutropenia
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 1994-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Chandler Dale, Study Chair — University of Washington
Locations (10):
- United States (5):
  - Dana-Farber/Boston Children¹s Cancer and Blood Disorders Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - St. Joseph's Children's Hospital, Paterson, New Jersey
  - University of Washington School of Medicine, Seattle, Washington
- Monash University, Melbourne, Victoria, Australia
- Canada (2):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Hospital for Sick Children, Toronto, Ontario
- Medizinische Hochschule Hannover, Hanover, Germany
- Leeds Teaching Hospitals, Yorkshire Regional Centre for Paediatric Oncology & Haematology, Leeds, England, United Kingdom

REFERENCES:
- [Background] Dale DC, Bonilla MA, Boxer L, et al.: Development of AML/MDS in a subset of patients (PTS) with severe chronic neutropenia (SCN). Blood 84(10 suppl 1): 518a, 1994.
- [Background] Guerra J, Withers DA, Boxer LM. Myb binding sites mediate negative regulation of c-myb expression in T-cell lines. Blood. 1995 Sep 1;86(5):1873-80. PMID 7655015
- [Background] Welte K, Dale D. Pathophysiology and treatment of severe chronic neutropenia. Ann Hematol. 1996 Apr;72(4):158-65. doi: 10.1007/s002770050156. PMID 8624368
- [Background] Kalra R, Dale D, Freedman M, Bonilla MA, Weinblatt M, Ganser A, Bowman P, Abish S, Priest J, Oseas RS, Olson K, Paderanga D, Shannon K. Monosomy 7 and activating RAS mutations accompany malignant transformation in patients with congenital neutropenia. Blood. 1995 Dec 15;86(12):4579-86. PMID 8541548